CLINICAL TRIAL: NCT02927938
Title: Leukemia Stem Cell Detection in Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated 7/23/2019 due to limited participation and testing challenges.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI-HEM-AML-SCD-001
Record Dates: First submitted 2016-09-29; First posted 2016-10-07 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Transplantation; Peripheral Blood Stem Cell Transplantation; Consolidation Chemotherapy; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Evaluable Cohort - Transplant Arm (Other): Other - Standard of Care Consolidation (HCT)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT); HMA-based induction subjects: Are candidates for (as determined by the investigator) and receive HCT
  Interventions: Procedure: Allogeneic HCT
- Evaluable Cohort - Consolidation Chemo Arm (Other): Other - Standard of Care Consolidation (cytarabine-based chemo)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT)
  Interventions: Drug: Consolidation chemotherapy
- Observational Cohort 1 (No Intervention): Enrolled subjects who do not achieve a CR to induction therapy, regardless of diagnostic phenotype. Following completion of induction therapy and remission bone marrow aspirate, if a subject is determined to not have achieved a complete remission to induction therapy, he or she would be included in observational cohort 1.
- Observational Cohort 2 (No Intervention): Enrolled subjects who achieve a CR to induction therapy but meet one or more of the following criteria:
  * Lack the immunophenotype of interest,
  * Cytarabine based induction subjects: Are not candidates for [as determined by the investigator (e.g. unfit or refusal)] and do not receive consolidation therapy (cytarabine-based chemotherapy or HCT)
  * HMA-based induction subjects: Are not candidates for [as determined by the investigator (e.g. unfit, lack of donor, refusal)] and do not receive HCT
  Final investigator determination of fit-ness can occur at any time until the start of consolidation therapy.
  HMA-based induction subjects will not receive consolidation cytarabine-based chemotherapy as part of the evaluable cohort if they do not receive HCT.

INTERVENTIONS:
Procedure: Allogeneic HCT — Allogeneic HCT
  Other Names: transplant, allo HCT, PBSCT, SCT, BMT
  Arms: Evaluable Cohort - Transplant Arm
Drug: Consolidation chemotherapy — Cytarabine-based consolidation chemotherapy
  Other Names: cytarabine, HiDAc, high dose cytarabine
  Arms: Evaluable Cohort - Consolidation Chemo Arm

SUMMARY:
Most patients with acute myeloid leukemia (AML) achieve complete remission (CR) following induction chemotherapy. However, a large majority subsequently relapse and succumb to the disease. Currently, cytogenetics and molecular aberrations are the best prognostic indicators; however, these factors cannot prognosticate accurately for individual patients. Overall, the majority of patients with favorable or intermediate-risk AML will experience relapse. Prognosis after relapse is dismal with a five-year overall survival rate of less than 10%. A leukemia stem cell (LSC) paradigm may explain this failure of CR to reliably translate into cure. This study is undertaken to determine whether the presence of LSCs has prognostic value as well as to determine whether the presence of LSCs has predictive value. This study has an observational component, whereby we intent evaluate whether the presence or absence of LSCs is prognostic. This study also has an interventional component in which it uses LSC status to determine whether favorable and intermediate risk AML patients in CR receive consolidation with chemotherapy or allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

1. Must have previously signed the specimen procurement protocol consent associated with the leukemia stem cell assay ("Step 1 informed consent") prior to starting AML therapy.
2. Age 18 years and older
3. New diagnosis of AML, other than APL, confirmed by bone marrow aspirate/biopsy and reviewed by an institutional hematopathologist
4. Completion of induction therapy, as defined by the Investigator and post-induction bone marrow biopsy.

Exclusion Criteria:

1. Any debilitating medical or psychiatric illness that would preclude ability to follow study procedures.
2. Indeterminate leukemia stem cell assay results at diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09; Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grunwald, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evaluable Cohort - Transplant Arm: Standard of Care Consolidation (HCT)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT); HMA-based induction subjects: Are candidates for (as determined by the investigator) and receive HCT
  Allogeneic HCT
- Evaluable Cohort - Consolidation Chemo Arm: Standard of Care Consolidation (cytarabine-based chemo)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT)
  Consolidation chemotherapy: Cytarabine-based consolidation chemotherapy
Period: Overall Study
Arm/Group | Evaluable Cohort - Transplant Arm | Evaluable Cohort - Consolidation Chemo Arm | Observational Cohort 1 | Observational Cohort 2
Started (Started/enrollment date is the date that the post-induction bone marrow aspirate was obtained.) | 1 | 6 | 4 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 6 | 4 | 7
Not completed — Death | 0 | 1 | 0 | 4
Not completed — Early Study Termination | 1 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Evaluable Cohort - Transplant Arm: Standard of Care Consolidation (HCT)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT); HMA-based induction subjects: Are candidates for (as determined by the investigator) and receive HCT
  Consolidation chemotherapy: Cytarabine-based consolidation chemotherapy
- Total: Total of all reporting groups
Arm/Group | Evaluable Cohort - Transplant Arm | Evaluable Cohort - Consolidation Chemo Arm | Observational Cohort 1 | Observational Cohort 2 | Total
Number analyzed (Participants) | 1 | 6 | 4 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants] — Age at date of consent
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 1 | 5 | 4 | 6 | 16
    >=65 years | 0 | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at date of consent
  years | 35.0 (NA) — No standard deviation can be calculated as there is only one subject in this group | 44.3 (14.7) | 51.0 (14.5) | 46.3 (15.6) | 46.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4 | 8
  Male | 1 | 4 | 2 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 6 | 4 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 2 | 7
  White | 1 | 4 | 1 | 4 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 6 | 4 | 7 | 18
AML Risk Level (prior to induction) [Count of Participants; unit: Participants] — AML risk level is determined from bone marrow biopsy performed at AML diagnosis
  * Unfavorable: complex karyotype (≥3 clonal chromosomal abnormalities); monosomal karyotype; -5 or 5q-; -7 or 7q-; 11q23 [non t(9;11)]; inv(3) or t(3;3); t(6;9); t(9;22); normal cytogenetics with FLT3-ITD mutation, therapy-related AML, or AML from myelodysplastic syndrome or myeloproliferative neoplasm
  * Favorable: t(8;21); inv(16) and/or t(16;16), or normal cytogenetics with NPM1 and/or dual CEBPA mutations without FLT3-ITD mutation
  * Intermediate: not meeting favorable or unfavorable definitions.
  Participants
    Favorable Risk | 0 | 6 | 1 | 4 | 11
    Intermediate Risk | 0 | 0 | 2 | 1 | 3
    Unfavorable Risk | 1 | 0 | 1 | 2 | 4
Immunophenotype at LSC0 [Count of Participants; unit: Participants] — LSC0: Diagnostic bone marrow sample or peripheral blood sample that the leukemia stem cell assay is performed on. LSC0 occurs prior to induction therapy for diagnostic purposes and identifies the subject's immunophenotype at diagnosis.
  Participants
    CD34- | 0 | 0 | 1 | 5 | 6
    CD34+CD38-ALDH(int) | 1 | 6 | 3 | 1 | 11
    CD34+CD38-ALDH(high) | 0 | 0 | 0 | 1 | 1
LSC0 Status (prior to induction) [Count of Participants; unit: Participants] — LSC0: Diagnostic bone marrow sample or peripheral blood sample that the leukemia stem cell assay is performed on. LSC0 occurs prior to induction therapy for diagnostic purposes.
  Participants
    Leukemia Stem Cells Detected | 1 | 6 | 3 | 1 | 11
    Leukemia Stem Cells Not Detected | 0 | 0 | 1 | 6 | 7
Deletion 5 or 5q [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 6 | 4 | 7 | 18
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
Deletion 7 or 7q [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 6 | 4 | 7 | 18
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
KNMT2A [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 6 | 4 | 7 | 18
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
inv(3) or t(3;3) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 5 | 4 | 7 | 17
    Uninterpretable results | 0 | 1 | 0 | 0 | 1
t(6;9) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 5 | 4 | 7 | 17
    Uninterpretable results | 0 | 1 | 0 | 0 | 1
t(9;22) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 5 | 4 | 7 | 17
    Uninterpretable results | 0 | 1 | 0 | 0 | 1
t(8;21) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 2 | 0 | 1 | 3
    Negative | 1 | 4 | 4 | 6 | 15
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
inv(16 or t(16;16) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 2 | 0 | 0 | 2
    Negative | 1 | 4 | 4 | 7 | 16
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
Plus 8 [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 6 | 4 | 7 | 18
    Uninterpretable results | 0 | 0 | 0 | 0 | 0
Plus 21 [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 5 | 4 | 7 | 17
    Uninterpretable results | 0 | 1 | 0 | 0 | 1
t(9;11) [Count of Participants; unit: Participants] — Cytogenetic and/or molecular abnormalities determined at diagnosis (LSC0 time point)
  Participants
    Positive | 0 | 0 | 0 | 0 | 0
    Negative | 1 | 5 | 4 | 7 | 17
    Uninterpretable results | 0 | 1 | 0 | 0 | 1
LSC1 Status (post induction, at enrollment) [Count of Participants; unit: Participants] — LSC1: Bone marrow sample that the post-induction leukemia stem cell (LSC) assay is performed on. LSC1 occurs following induction therapy and at the time of complete remission assessment (End of Induction visit).
  Participants
    Leukemia Stem Cells Detected | 0 | 0 | 1 | 1 | 2
    Leukemia Stem Cells Not Detected | 0 | 6 | 2 | 4 | 12
    Indeterminate/Unknown Results | 1 | 0 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Relapse Free Survival (RFS)
Description: Comparison of 2 year RFS in patient with detectable LSCs in the marrow at the end of consolidation to the 2 year RFS of patients without detectable LSCs. IWG Criteria (Cheson 2003) was utilized to classify relapse, with relapse defined as ≥ 5% blasts in the marrow or peripheral blood, extramedullary disease, or disease presence determined by a physician upon clinical assessment.
Time Frame: 2 years
Population: The primary efficacy analyses will be conducted on the subset of subjects who were included in the evaluable cohort (HCT or chemo treatment arm) and who also had a successful/interpretable end of consolidation eLSC assay. This excludes subjects in OC1 and 2, as they did not achieve CR to induction or did not have the immunophenotype of interest.
Measure: Count of Participants; unit: Participants
Groups:
- eLSC+ (Evaluable Cohort): Of the subjects enrolled in the evaluable cohort (either allo HCT or consolidation chemotherapy), those who had leukemia stem cells detected post-consolidation. Note, eLSC indicates the time point after consolidation.
- eLSC- (Evaluable Cohort): Of the subjects enrolled in the evaluable cohort (either allo HCT or consolidation chemotherapy), those who had leukemia stem cells not detected post-consolidation. Note, eLSC indicates the time point after consolidation.
Arm/Group | eLSC+ (Evaluable Cohort) | eLSC- (Evaluable Cohort)
Number analyzed (Participants) | 0 | 5
Participants |  | NA — Study terminated early, with immature outcome data. There was not enough follow up to determine 2-year RFS status for these subjects prior to study termination.

ADVERSE EVENTS:
Time Frame: Graft Versus Host Disease (GVHD) events were collected from the time of consolidation HCT through long term follow-up (up to approximately 5 years). - Acute GVHD: Confirmed GVHD within 100 days of HCT. - Chronic GVHD: Confirmed GVHD 100 days or more after HCT.
Description: Both cytarabine-based consolidation chemo and HCT are considered standard of care for this disease population. With the exception of GVHD, an event of clinical interest, adverse events experienced by the subjects were not recorded in the dataset or included in the safety analysis. Each occurrence of GVHD, in evaluable subjects who received HCT, was graded by the investigator according to accepted institutional practice: CIBMTR grading for Acute GVHD; NIH Consensus criteria for Chronic GVHD.
Groups:
- Evaluable Cohort - Transplant Arm: Standard of Care Consolidation (HCT)
  Enrolled subjects that will contribute to the population of subjects who are evaluable for the primary and secondary objectives. This will not include any subjects who end up in either observational cohort. To be included in the evaluable cohort, the subject must meet the following requirements:
  1. Complete remission (CR1) from standard cytarabine or HMA-based induction therapy per standard clinical criteria (Cheson Criteria)
  2. Have confirmed presence of CD34+CD38-ALDHint population by flow cytometry at the diagnostic LSC assay (LSC0)
  3. Cytarabine-based induction subjects: Are candidates for (as determined by the investigator) and receive consolidation therapy (cytarabine-based chemotherapy or HCT); HMA-based induction subjects: Are candidates for (as determined by the investigator) and receive HCT
  Allogeneic HCT: Allogeneic HCT
Arm/Group | Evaluable Cohort - Transplant Arm | Evaluable Cohort - Consolidation Chemo Arm | Observational Cohort 1 | Observational Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/6 | 0/4 | 4/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/6 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/1 | 0/6 | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT02927938/Prot_SAP_000.pdf